CLINICAL TRIAL: NCT01207128
Title: A Phase II Randomized, Double Blind, Placebo-controlled, Trial of Combination Antifungal Therapy (Voriconazole Plus Micafungin vs. Voriconazole Plus Placebo Equivalent) in the Treatment of Invasive Aspergillosis (IA) in Patients With Hematological Cancer
Brief Title: Trial of Combination Antifungal Therapy (Vori+Mica vs. Vori+Placebo) in Invasive Aspergillosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: None enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UARK 2010-14
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole; Micafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voriconazole, Micafungin (Active Comparator): Patients will receive either IV micafungin 100 mg or placebo equivalent daily. Intravenous (IV) Voriconazole will be administered at a loading dose of 6 mg/kg every 12 hours for the first 24 hours followed by a maintenance dose of 4 mg/kg every 12 hours. Patients may be switched to oral voriconazole 200 mg BID provided aspergillosis response is achieved and gastrointestinal functions are intact.
  Interventions: Drug: Voriconazole, micafungin
- Voriconazole+Micafungin or Voriconazole+Placebo (No Intervention): Voriconazole+Micafungin or Voriconazole+Placebo

INTERVENTIONS:
Drug: Voriconazole, micafungin — Patients will receive either IV micafungin 100 mg or placebo equivalent daily. Intravenous (IV)Voriconazole will be administered at a loading dose of 6 mg/kg every 12 hours for the first 24 hours followed by a maintenance dose of 4 mg/kg every 12 hours. Patients may be switched to oral voriconazole 200 mg BID provided aspergillosis response is achieved and gastrointestinal functions are intact.
  Arms: Voriconazole, Micafungin

SUMMARY:
The purpose of this study is to evaluate the therapeutic effectiveness of combination antifungal therapy (CAT) of voriconazole plus micafungin versus voriconazole plus placebo equivalent as primary therapy for invasive aspergillosis (IA) in patients with hematological cancer.

DETAILED DESCRIPTION:
Patients will receive either IV micafungin 100 mg or placebo equivalent daily. Intravenous (IV)Voriconazole will be administered at a loading dose of 6 mg/kg every 12 hours for the first 24 hours followed by a maintenance dose of 4 mg/kg every 12 hours. Patients may be switched to oral voriconazole 200 mg BID provided aspergillosis response is achieved and gastrointestinal functions are intact.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legally authorized representative has signed an informed consent/assent.

   Assent will be obtained as required by the UAMS IRB.
2. The patient has a diagnosis of proven or probable invasive aspergillosis and with positive Aspergillus GM index (≥0.5 ng/ml) provide the patient is not receiving antibiotics, such as piperacillin-tazobactam, that are known to cause false positive GMI
3. The patient is 18 years of age or older.

Exclusion Criteria:

1. The patient is being treated with an unlicensed investigational drug for aspergillosis.
2. The patient has been administered an antifungal agent (voriconazole, itraconazole, posaconazole, caspofungin, micafungin, anidulafungin, amphotericin B, or lipid formulation of amphotericin B) for > 7 days immediately prior to randomization for treatment of the Probable, or Proven invasive aspergillosis for which the patient is being enrolled.
3. Patient has invasive aspergillosis but with negative Aspergillus GM index.
4. The patient is pregnant or lactating. If the patient is female and of childbearing potential, the patient must have a negative pregnancy test and avoid becoming pregnant while receiving study drug. A pregnancy test should be performed within 14 days prior to the first dose of study drug.
5. The patient has alkaline phosphatase, ALT, AST or total bilirubin greater than five times the upper limit of normal.
6. The patient has hepatic cirrhosis.
7. Patients with creatinine > 3 will be enrolled only if able to receive oral voriconazole (specify oral loading dose is 6 mg/kg PO Q 12 hours for 24 hours) then oral maintenance 200 mg PO q 12 hours).
8. The patient is on artificial ventilation, and unlikely to be extubated within 24 hours of study entry.
9. The patient has a history of allergy, hypersensitivity, or any serious reaction to the azole or echinocandin class of antifungal agents.
10. The patient has previously enrolled into this study.
11. The patient has a concomitant medical condition, which in the opinion of the Investigator may create an unacceptable additional risk.
12. The patient has an active microbiologically-documented deep infection due to a non-Aspergillus mold.
13. The patient has a life expectancy of less than seven days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Response | maximum 6 weeks
  Response is defined as normalization of the serum Aspergillus galactomannan index (GMI)values (first normal GMI value is considered day of response).

CONTACTS AND LOCATIONS:
Overall Officials: Elias Anaissie, MD, Study Chair — University of Arkansas
Locations (2):
- United States (2):
  - UAMS, Little Rock, Arkansas
  - University of Arkansas, Little Rock, Arkansas